CLINICAL TRIAL: NCT05539963
Title: A Multi-center, Randomized, Controlled Feasibility Trial of STIMULAN VG and Debridement With an Abbreviated Course of Systemic Antibiotics to Debridement and a Full Course of Systemic Antibiotics for the Treatment of Diabetic Foot Osteomyelitis
Brief Title: A Feasibility Trial to Investigate the Safety and Between-group Effect Size of STIMULAN VG and Standard of Care (SoC) in Participants With Diabetic Foot Osteomyelitis
Acronym: BLADE-VG2
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Biocomposites Ltd (Industry)
Collaborators: MCRA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 254915
Expanded Access: NCT06808568 (Available)
Record Dates: First submitted 2022-09-12; First posted 2022-09-14 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Diabetic Foot Osteomyelitis
Keywords: feasibility; between-group effect size; surgical debridement; systemic antibiotic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- STIMULAN VG (Experimental): Participants will receive STIMULAN VG on Day 1 following surgical debridement. Systemic antibiotics for 3 days ± 2 days following the debridement surgery.
  Interventions: Drug: STIMULAN VG; Drug: Systemic Antibiotics
- Standard of Care (Active Comparator): Participants will receive Systemic antibiotics for 4-6 weeks following the debridement surgery.
  Interventions: Drug: Systemic Antibiotics

INTERVENTIONS:
Drug: STIMULAN VG — Participants will receive STIMULAN VG via implantation during debridement surgery on Day 1.
  Arms: STIMULAN VG
Drug: Systemic Antibiotics — Participants will receive Antibiotics per site-specific requirements.

SUMMARY:
The purpose of this trial is to evaluate the safety and between-group effect size of STIMULAN VG compared to SoC treatment in patients with diabetic foot osteomyelitis (DFO).

DETAILED DESCRIPTION:
This trial is an open-label, multi-center, randomized, controlled feasibility trial.

All participants will undergo surgical debridement and receive either STIMULAN VG and an abbreviated course of systemic antibiotic therapy (3 days ±2 days) or a full course (4-6 weeks) of systemic antibiotic therapy.

The total duration of study is Approximately 55 weeks.

ELIGIBILITY:
Inclusion Criteria:

Participants are eligible to be included in the trial only if all of the following criteria apply:

1. Participant must be ≥18 years of age inclusive, at the time of signing the informed consent
2. Participant has a current diagnosis and is being treated for diabetes mellitus, type 1 or type 2
3. Participant who has confirmed presence of DFO (to include all bones below the ankle including the talus and calcaneum) as evidenced by at least 3 out of 5 of the following:

   1. Positive PTB test
   2. Presence of draining sinus presumed to be from underlying bone
   3. Plain X-ray or MRI scan highly suggestive of or most compatible with osteomyelitis
   4. Ulcer present for greater than 30 days
   5. Substantially elevated serum marker for inflammation (e.g. ESR >70 mm/hr and C-reactive protein >14mg/L or at least 40% higher than upper limits of normal value used at the investigational site)
4. Participant who requires surgical debridement OR Participant requiring amputation and/or resection where residual osteomyelitis remains that necessitates further surgical debridement
5. All genders are eligible to participate if they are not pregnant, not breastfeeding, are not of childbearing potential or they agree to follow contraceptive guidance
6. Subject or legal authorized representative able to provide, voluntary, signed and dated informed consent prior to any study related procedures

Exclusion criteria:

Participants are excluded from the trial if any of the following criteria apply:

1. Osteomyelitis in any location other than the foot (i.e. excluding any bones located proximal to the foot)
2. Osteomyelitis of the distal phalanx (toe tip) of the great toe or lesser toes
3. Charcot foot or other deformities where the investigator believes adequate offloading is not possible
4. Severe diabetic foot infection (grade 4) in accordance to IDSA/IWGDF criteria (Appendix 6)
5. Moderate to severe reduction in renal function, defined as estimated glomerular filtration rate (eGFR) of < 30.0 ml/min/1.73 m2 (Formula for calculating eGFR: 2021 CKD-EPI Creatinine).
6. Significant peripheral arterial disease:

   * Ankle brachial index ≤ 0.7 mm Hg OR
   * toe pressure ≤ 40 mm Hg OR
   * transcutaneous oximetry ≤ 40 mm Hg
7. Hemoglobin A1c (HbA1c) > 12%
8. Contra-indication or inability to undergo an MRI scan
9. Malignancy that might affect trial interpretation of outcomes or the participant's ability to complete the trial
10. Participant who is severely immunocompromised or has received high dose corticosteroids (>10 mg prednisone (or corticosteroid equivalent) for more than 14 consecutive days within the 90 days prior to informed consent)
11. Any conditions with known hypercalcemia (> 10.3 mg/dl) or posing a significant risk for developing hypercalcemia (i.e., Hyperparathyroidism)
12. Patients with active COVID-19 will be excluded from enrollment until they are able to undergo the surgical procedure
13. Current or recent history (within last 2 years) of active substance abuse (e.g. recreational drugs, narcotics, or alcohol) that, in the judgment of the investigator, may compromise the ability of the trial participant to adhere to the trial conduct and procedures
14. Previous history of adverse incidents, allergy or contra indications (e.g. Myathesia Gravis) to any component of the investigational product, such as calcium sulfate, glycopeptide antibiotics (vancomycin), or aminoglycoside antibiotics (gentamicin)
15. Concurrent involvement in a trial of another investigational product
16. The Investigator believes trial participation may compromise safety of the participant or the results of the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2023-01-23 (Actual); Primary Completion 2025-06-20 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants with confirmed absence of clinical signs of osteomyelitis or surgical infection at the index site | Week 24
  Confirmed absence of clinical signs of osteomyelitis or surgical site infection at the index site will be evidenced by Negative Probe to Bone Test (PTB), absence of draining sinus presumed to be from underlying bone and MRI scan at Week 24.
Number of participants with no clinical need for further antibiotic therapy for infection at the index site | Week 24
  Need for further antibiotic therapy for infection at the index site will be assessed at Week 24.
Number of participants with no clinical need for further additional surgical procedure or debridement to treat infection at the index site | Week 24
  Need for further additional surgical procedure or debridement to treat infection at the index site will be assessed at Week 24.

SECONDARY OUTCOMES:
Ulcer healing per the University of Texas (UT) Staging System for Diabetic Foot Ulcers | Week 12
  The Investigator will assess the ulcer for healing using the UT Staging System for Diabetic Foot Ulcers which grades DFUs by grade (0, I, II, III) and stage (A, B, C, D), depending on the presence or absence of infection and ischemia. The grades are referred to as follows: grade 0 (pre-or post-ulcerative site that has healed), grade 1 (superficial ulcer not involving tendon, capsule, or bone), and grade 2 (ulcer penetrating to tendon or capsule), and grade 3 (ulcer penetrating bone or joint). The patient will be scored based on Grade score and stage score together. Grade 0, stage A considered being low severity, and Grade 3, stage D considered to be more severe.
Number of participants with occurrence of reinfection at the index site | Week 52
  Number of participants with the occurrence of reinfection at the index site will be assessed via PTB, absence of draining sinus presumed to be from underlying bone and MRI at Week 52.
Number of participants with no clinical need for further antibiotic therapy for infection at the index site | Week 52
  Need for further antibiotic therapy for infection at the index site will be assessed at Week 52.
Number of participants with no clinical need for further additional surgical procedure or debridement to treat infection at the index site | Week 52
  Need for further additional surgical procedure or debridement to treat infection at the index site will be assessed at Week 52.
Relative change from baseline in Cardiff Wound Impact Schedule (CWIS) quality of life assessment | Week 24
  The CWIS is designed and validated to specifically assess the quality of life (QoL) of subjects with chronic wounds (leg ulcers and diabetic foot ulcers (DFU)). This questionnaire contains 47 items divided into four scales: demographic and clinical characteristics (3 items), global health-related quality of life (HRQoL) (1 item), satisfaction with HRQoL (1 item) and impact of the wound on lifestyle. This last scale includes 3 domains: social life (14 items in total, 7 related to stress and 7 to experience), wellbeing (7 items), and physical symptoms and everyday living (24 items in total, 12 related to stress and 12 to experience). All three domains are scored on a 5-point scale, from "not at all" to "always". Thus, the total score includes the patient's perception of the experience and the associated stress. The final score ranges from 0 (poorer QoL) to 100 points (higher QoL) where a high score indicates a positive rating
Number of participants with adverse events | Week 52
  The number of participants with adverse events will be assessed.
Number of participants discontinuing therapy prematurely due to a treatment related event | Week 52
  The number of participants discontinuing therapy prematurely due to a treatment-related event will be assessed during the course of the trial and recorded on the participants electronic case report form (eCRF).
Number of hospitalizations/re-hospitalizations as a result of treatment for osteomyelitis or ulceration at the index site | Week 52
  The number of hospitalizations/re-hospitalizations as a result of treatment for osteomyelitis will be assessed during the course of the trial and recorded on the participants eCRF.
Number of participants undergoing amputation at the index site | Week 52
  The number of participants undergoing amputation at the index site will be assessed during the course of the trial and recorded on the participants eCRF.
Number of systemic antibiotic free days since trial surgery | Week 52
  The total number of days from Day 1 to week 24 without the use of antibiotics.

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - Titan Clinical Research, Mesa, Arizona
  - Axsendo Clinical Research, Phoenix, Arizona
  - Perseverance Research Center, LLC, Scottsdale, Arizona
  - Advanced Footcare LLC, Scottsdale, Arizona
  - NEA Baptist Clinic, Jonesboro, Arkansas
  - Viable Clinical Research, Henderson, Nevada
  - Equitable Health Partners - NJ, Mountainside, New Jersey
  - Mount Sinai West, New York, New York
  - UNC School Medicine, Chapel Hill, North Carolina
  - Seaside Clinical Research Institute, Wilmington, North Carolina

IPD SHARING:
Plan to Share IPD: No